CLINICAL TRIAL: NCT05265559
Title: Multicenter Prospective Clinical Trial of Partial Ceramic Posterior Restorations Using Immediate Dentin Sealing - The Infuence of Operator Factors on Success and Survival
Brief Title: Influence of Operator Factors on Succes and Survival of Indirect Restorations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201800678
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Partial Indirect Restoration; Clinical Study; Adhesion; Immediate Dentin Sealing; Posterior Region; Operator Factors
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Partial Indirect Restoration — Dental restorative treatment

SUMMARY:
Background: Nowadays, tissue preserving, aesthetically high-quality and sustainable dentistry is more and more becoming the standard way of treatment. To reach those standards, one of the treatment options is applying a partial indirect restoration made by glass ceramics using immediate dental sealing (IDS). Using IDS, a protocol is followed to applicate a dentin bonding agent to freshly cut dentin when it is exposed during tooth preparation for indirect restorations (inlays/onlays, crowns). The preparation made for partial restorations is minimal invasive. Glass ceramic restorations have very high survival rates (90 to 100% after five years) (Morimoto et al., 2016) and glass ceramic mimics the color and structure of the tooth very well.

This kind of treatment is gaining interest and increasingly applied however little information is available on the long-term effects when multiple general practitioners apply these restorations.

Objectives: The main goal of this study is to evaluate partial posterior ceramic restorations with the application of an immediate dentin sealing (IDS) performed by various practitioners.

Study design and population:

Twenty dental practitioners, who followed a course on making ceramic partial restorations using IDS, will be asked to include patients for this study. The dental practitioners are being asked to share their data (occlusal light photo's, impression and x-rays) of twenty-five restorations they make after having the course. Restorations of individuals with a minimum age of 18 will be included. The information from pictures and impressions will be evaluated.

Items to evaluate

The practitioners will be interviewed to get to know in what circumstances they do their treatment. Items that are discussed are:

* using rubber dam;
* using magnification by means of loupes/microscope;
* scheduled time for the treatment;
* number of restorations after following the course.

Initial data (gathered directly after treatment) will be evaluated looking at:

* surface of preparation after IDS;
* size of the prepared surface;
* color.

Follow up data will be evaluated looking at:

* tooth extraction
* fracture restoration
* fracture tooth
* secondairy caries
* de-bonding
* endodontic problems

Outcome: Failures (fracture, de-bonding, secondairy cariës, endodontic problems) are the main outcome measurements.

Description and estimation of the load and risk for the subjects:

No extra intervention is performed. The dental practitioners will provide their data (i.e. impressions, occlusal light photo's) and these will be evaluated by the researchers. Follow up data will be gathered from X-rays already made for periodical oral examination (taking the caries risk into account). Summarizing, there is no extra load or risk for the patients.

Studie design Prospective practice-based research, multicenter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Adults

Exclusion Criteria:

* Periodontal unstable situation
* Endodontic unstable situation
* Allergies for one or more of the used products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ten different dentists will ask patients (who have been indicated and agreed to have an indirect restoration) if they would like to be part of this study. Taking possible drop-out into account, the practitioners are asked to include twenty patients each (total n=200).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Survival and Succes | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided